CLINICAL TRIAL: NCT03960762
Title: COMPARISON OF ERECTOR SPINAE PLANE BLOCK AND SERRATUS ANTERIOR PLANE BLOCK FOR POSTOPERATİVE ANALGESIA MANAGEMENT FOLLOWING VIDEO ASSISTED THORACIC SURGERY
Brief Title: Erector Spinae Plane Block or Serratus Anterior Plane (SAP) Block Following Video Assisted Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Primary researcher, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Mega
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Lung Diseases
Keywords: Video assisted thoracic surgery; Postoperative pain management; Erector spina plane block; Serratus anterior plane block
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Intervention Model Description: Fifty patients aged 18-65 years old with American Society of Anesthesiologists (ASA) classification I-II and scheduled for VATS under general anesthesia will be included in the study. Patients with a history of bleeding diathesis, receiving anticoagulant treatment, known local anesthetics and opioid allergy, infection of the skin at the site of the needle puncture, pregnancy or lactation, and patients who do not accept the procedure will be excluded from the study. Randomization will be achieved using a randomizing computer program. Patients will be randomly divided into two groups (Group A = ESP group, Group B = SAP group) including 25 patients each, before entering the operating room.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcomes Assessor and participant will be blinded to the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A = ESP group (Active Comparator): ESP block (Group ESP) will be performed in the preoperative block room. Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. The PCA device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol included 20 mcg bolus without infusion dose, 20 min lockout time and 4 hour limit.
  Interventions: Other: ESP block (Group ESP)
- Group B = SAP group (Active Comparator): SAP block (Group SAP) will be performed in the preoperative block room. Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. The PCA device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol included 20 mcg bolus without infusion dose, 20 min lockout time and 4 hour limit.
  Interventions: Other: SAP block (Group SAP)

INTERVENTIONS:
Other: ESP block (Group ESP) — In group A, ESP block will be performed. US probe will be placed longitudinally 2-3 cm lateral to the T5 transverse process. From superior to inferior, three muscles will be visualized on the hyperechoic transverse process; trapezius (upper), rhomboideus major (middle), erector spinae (lower). The block needle will be inserted cranio caudal direction and then for correction of the needle 5 ml saline will be injected deep into the erector spina muscle fascia. Following confirmation of the correct position of the needle 20 ml %0.25 bupivacaine will be administered for block
  Arms: Group A = ESP group
Other: SAP block (Group SAP) — In group B, after lateral positioning, US probe will be placed in a sagittal plane over the midclavicular region of the thoracic cage. Then the 7th rib will be identified in the midaxillary line, followed by the identification of the following muscles overlying the 6th rib: the latissimus dorsi (superficial and posterior), teres major (superior), and serratus muscle (deep and inferior). The needle will be inserted in-plane with respect to the ultrasound probe targeting the plane superficial to the serratus anterior muscle. 5 ml saline will be enjected for correction. Following confirmation of the correct position of the needle 20 ml %0.25 bupivacaine will be administered for block.
  Arms: Group B = SAP group

SUMMARY:
Video assisted thoracic surgery (VATS) has recently been evaluated as the standard surgical procedure for lung surgery. Although VATS is less painful than thoracotomy, patients may feel severe pain during the first hours at postoperative period. Analgesia management is very important for these patients in postoperative period since insufficient analgesia can cause pulmonary complications such as atelectasis, pneumonia and increased oxygen consumption. The ultrasound (US) guided erector spina plane (ESP) block is a novel interfacial plan block defined by Forero et al. at 2016. ESP block provides thoracic analgesia at T5 level and abdominal analgesia at T7-9 level. Visualization of sonoanatomy with US is easy, and the spread of local anesthesic agents can be easily seen under the erector spinae muscle. Thus, analgesia occurs in several dermatomes with cephalad-caudad way. US-guided serratus anterior plane (SAP) block provides effective analgesia in anterior, posterior and lateral dermatomes of thorax. It has been reported that SAP block provides effective postoperative pain management following thoracotomy, breast surgery and VATS. There is no clinical randomized study evaluating the efficacy of ESP block and SAP block following VATS in the literature.

DETAILED DESCRIPTION:
Video assisted thoracic surgery (VATS) has recently been evaluated as the standard surgical procedure for lung surgery. The advantages of VATS procedures compared with open thoracotomy are rapid recovery, short hospital stay and low complication risk. Although VATS is less painful than thoracotomy, patients may feel severe pain during the first hours at postoperative period. Analgesia management is very important for these patients in postoperative period since insufficient analgesia can cause pulmonary complications such as atelectasis, pneumonia and increased oxygen consumption.

The ultrasound (US) guided erector spina plane (ESP) block is a novel interfacial plan block defined by Forero et al. at 2016. ESP block provides thoracic analgesia at T5 level and abdominal analgesia at T7-9 level. The ESP block contains a local anesthetic injection into the deep fascia of erector spinae. This area is away from the pleural and neurological structures and thus minimizes the risk of complications due to injury. Visualization of sonoanatomy with US is easy, and the spread of local anesthesic agents can be easily seen under the erector spinae muscle. Thus, analgesia occurs in several dermatomes with cephalad-caudad way. Cadaveric studies have shown that the injection spreads to the ventral and dorsal roots of the spinal nerves and creates sensory blockade in both posterior and anterolateral thorax. In the literature, it has been reported that ESP block provides effective analgesia after open heart surgery, breast surgery and ventral hernia repair in randomized controlled studies about ESP block efficiency for postoperative analgesia management. In some case series and case reports it has been reported that ESP block provides effective analgesia after thoracotomy and VATS. Furthermore, it has been reported that it provides effective analgesia in chronic and persistant pain syndromes of thorax.

US-guided serratus anterior plane (SAP) block is an interfascial plane block and was described by Blanco in 2013. A local anesthetic solution is performed into the fascial plane of serratus anterior muscle. It is easy to perform and has low complication rate because it is far away from the important neurological and vascular structures. The serratus anterior muscle may be seen easily with US guidance in the mid-axillary line. It provides effective analgesia in anterior, posterior and lateral dermatomes of thorax. It has been reported that SAP block provides effective postoperative pain management following thoracotomy, breast surgery and VATS. There is no clinical randomized study evaluating the efficacy of ESP block and SAP block following VATS in the literature.

The aim of this study is to compare US-guided ESP block and SAP block for postoperative analgesia management after VATS. The primary aim is to compare perioperative and postoperative opioid consumption and the secondary aim is to evaluate postoperative pain scores (VAS), adverse effects related with opioids (allergic reaction, nausea, vomiting) and complications due to blocks (pneumothorax, hematoma).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for VATS under general anesthesia

Exclusion Criteria:

* Bleeding diathesis
* Receiving anticoagulant treatment
* Known local anesthetics and opioid allergy
* Infection of the skin at the site of the needle puncture
* Pregnancy or lactation
* Patients who do not accept the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Opioid consumption by the patients at postoperative 24 hours period | Postoperative 24 hours
  Fentanyl using

SECONDARY OUTCOMES:
Postoperative pain scores | Postoperative 24 hours period
  Postoperative pain assessment will be performed using the VAS score (0 = no pain, 10 = the most severe pain felt). The VAS scores at rest and during cough will be recorded at postoperative 0, 2, 4, 8, 16 and 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Bahadir Ciftci, Asist.Prof, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared

REFERENCES:
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Gurkan Y, Aksu C, Kus A, Yorukoglu UH, Kilic CT. Ultrasound guided erector spinae plane block reduces postoperative opioid consumption following breast surgery: A randomized controlled study. J Clin Anesth. 2018 Nov;50:65-68. doi: 10.1016/j.jclinane.2018.06.033. Epub 2018 Jul 2. PMID 29980005
- [Background] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989
- [Background] Okmen K, Metin Okmen B. Evaluation of the effect of serratus anterior plane block for pain treatment after video-assisted thoracoscopic surgery. Anaesth Crit Care Pain Med. 2018 Aug;37(4):349-353. doi: 10.1016/j.accpm.2017.09.005. Epub 2017 Oct 12. PMID 29033355